CLINICAL TRIAL: NCT06560112
Title: An Exploratory, Multi-cohort Phase II Study of Combination Therapy With AK104 and AK112 for Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK104-221
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): AK104 q3w +Chemo
  Interventions: Drug: AK104; Drug: Chemotherapy
- Cohort 2 (Experimental): AK112 q3w +Chemo
  Interventions: Drug: AK112; Drug: Chemotherapy
- Cohort 3 (Experimental): AK112 q3w +AK104 q6w
  Interventions: Drug: AK104; Drug: AK112
- Cohort 4 (Experimental): AK112 q3w +AK104 q6w +Chemo
  Interventions: Drug: AK104; Drug: AK112; Drug: Chemotherapy

INTERVENTIONS:
Drug: AK104 — ivgtt
  Other Names: Cadonilimab
  Arms: Cohort 1; Cohort 3; Cohort 4
Drug: AK112 — ivgtt
  Other Names: Ivonescimab
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: Chemotherapy — ivgtt
  Other Names: Monotherapy Non-Platinum Chemotherapy chosen by the investigator
  Arms: Cohort 1; Cohort 2; Cohort 4

SUMMARY:
An Exploratory, Multi-cohort Phase II Study of Combination Therapy With AK104 and AK112 for Recurrent Ovarian Cancer

DETAILED DESCRIPTION:
This is a Phase 2, open label, multicohort, multicenter study designed to evaluate the efficacy and safety of combination therapy of AK104, AK112 and chemotherapy in recurrent ovarian cancer.

AK104 is a bispecific monoclonal antibody targeting both CTLA-4 and PD-1. AK112 is a bispecific monoclonal antibody targeting VEGF and PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. Signs the written informed consent form.
2. Female participants who are at least 18 years of age on the day of signing informed consent with.
3. ECOG of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Histologically diagnosed high-grade epithelial ovarian cancer (including high-grade serous, clear cell, G3 endometrioid) that has relapsed after platinum-containing standard chemotherapy.

   1. Recurrence of Platinum-sensitive (relapse ≥6 months after the end of platinum-containing therapy) who is not suitable for platinum-containing therapy after ≥ 3 lines of therapy;
   2. Recurrence of platinum resistance , ≤3 previous lines of therapy. Note: Ovarian cancer includes ovarian cancer, fallopian tube cancer and primary peritoneal cancer in this study, unless otherwise specified.
6. Has measurable disease based on RECIST v1.1 as determined by the site study team.
7. Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue.
8. Has adequate organ function.
9. All subjects of reproductive potential must agree to use an effective method of contraception, during and for 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Other pathological types such as mucinous cancer, low-grade serous carcinoma, carcinosarcoma, sex cord stromal cell tumor, etc.
2. Presence of central nervous system (CNS) metastases or carcinomatous meningitis.
3. Subjects with uncontrollable pleural, pericardial, or peritoneal effusion requiring repeated drainage.
4. Patients with other active malignancies within 3 years prior to randomization.
5. Received systemic anti-tumor therapy within 3 weeks prior to randomization.
6. Any prior treatments targeting the mechanism of tumor immunity.
7. Major surgical treatment, open biopsy or significant trauma within 4 weeks prior to randomization; or elective major surgical treatment required during the study.
8. Active or potentially recurrent autoimmune disease.
9. Subjects who require systemic treatment with glucocorticoid (> 10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to randomization.
10. Use of live vaccines within 4 weeks prior to randomization.
11. Known primary or secondary immunodeficiencies, including testing positive for human immunodeficiency virus (HIV) antibodies.
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Known history of interstitial lung disease or non-infectious pneumonitis.
14. Serious infections requiring hospitalization.
15. Presence of active infection requiring systemic therapy.
16. Subjects with active hepatitis B and active viral hepatitis C.
17. Active or documented inflammatory bowel diseases, active diverticulitis.
18. Patients with clinically significant cardio-cerebrovascular disease.
19. Unresolved toxicities from prior anticancer therapy.
20. History of severe hypersensitivity reactions to other mAbs.
21. Pregnant or lactating women.
22. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug.
23. Exclusion Criteria for Chemotherapy-Related Cohorts (Cohorts 1,2,4): Known contraindications or allergy to PLD, paclitaxel or topotecan.
24. Exclusion Criteria for AK112-Related Cohorts (Cohorts 2,3,4): Known contraindications or allergy to any component of VEGF mABs or any medical conditions that affect the safety of AK112.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by investigator | Up to 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
progression-free survival (PFS) assessed by investigator per RECIST v1.1 | Up to 2 years
  PFS is defined as the time from the date of first dosing till the first documented disease progression (Per RECIST v1.1 assessed by the investigator) or death due to any cause, whichever occurs first.
duration of Response (DOR) assessed by investigator per RECIST v1.1 | Up to 2 years
  DOR means time measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Time to Response (TTR) assessed by investigator per RECIST v1.1 | Up to 2 years
  TTR refers to Time to Response.
Overall Survival(OS) | Up to 2 years
  OS is defined as the time from randomization or first dosing to death due to any cause.
Number of participants with adverse event (AE) | Up to 2 years
  The number of participants experiencing an Adverse Event (AE) and the severity of AEs will be assessed. AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No